CLINICAL TRIAL: NCT02340247
Title: Effects of Ursodeoxycholic Acid and Chenodeoxycholic Acid on GLP-1 Secretion After Roux-en-Y Gastric Bypass
Brief Title: Effects of Bile Acids on GLP-1 Secretion After Roux-en-Y Gastric Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Maria Saur Svane, MD, Hvidovre University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SN-GALDE-14
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Severe Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Water; Ursodeoxycholic Acid; Chenodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Experimental): 150mL water
  Interventions: Other: Water
- Ursodeoxycholic acid (Experimental): Ursodeoxycholic acid (750mg) dissolved in 150mL water
  Interventions: Drug: Ursodeoxycholic Acid
- Chenodeoxycholic acid (Experimental): Chenodeoxycholic acid (1250mg) dissolved in 150mL water
  Interventions: Drug: Chenodeoxycholic Acid

INTERVENTIONS:
Other: Water
  Arms: Placebo
Drug: Ursodeoxycholic Acid
  Arms: Ursodeoxycholic acid
Drug: Chenodeoxycholic Acid
  Arms: Chenodeoxycholic acid

SUMMARY:
The purpose of this study is to examine the effects of bile acids on GLP-1 secretion after Roux-en-Y gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated RYGB performed minimum 3 months prior to the study.
* Fasting plasma glucose < 7.0mM, HbA1c < 48mmol/mol 3 months after RYGB.

Exclusion Criteria:

* Fasting plasma glucose > 7.0mM, HbA1c > 48mmol/mol 3 months after RYGB.
* Dysregulated hypothyroidism, use of antithyroid treatment.
* Late diabetic complications as retinopathy, renal insufficiency, neuropathy or previous pancreatitis.
* Complications to RYGB: Documented reactive hypoglycaemia, severe dumping (vomiting, diarrhea, severe abdominal pain after food intake).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
GLP-1 secretion (evaluated by iAUC) | Baseline, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180

SECONDARY OUTCOMES:
C-peptide secretion (evaluated by iAUC) | Baseline, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180
PYY secretion (evaluated by iAUC) | Baseline, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180
Glucagon secretion (evaluated by iAUC) | Baseline, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180
GIP secretion (evaluated by iAUC) | Baseline, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180
CCK secretion (evaluated by iAUC) | Baseline, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180
Gherlin secretion (evaluated by iAUC) | Baseline, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180
Changes in bile acids/FGF-19 | Baseline, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180
TSH/T3/T4 | 0, 60, 120, 180
Appetite measurements (VAS-score) | Baseline, 30, 60, 120, 180

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark